CLINICAL TRIAL: NCT07257770
Title: Evaluating the Effect of a Medical Device Based on Inositol in Improving Breast Pain
Brief Title: Local Treatment of Breast Pain Based on the Daily Use of a Topical Gel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INO-BREAST
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Mastalgia
Keywords: inositol; breast pain; mastalgia
MeSH Terms: conditions — Mastodynia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No treatment, clinical follow up
- treatment inositol (Experimental): daily administration of the gel
  Interventions: Device: inositol

INTERVENTIONS:
Device: inositol — Topical application of a medical device based on inositol
  Arms: treatment inositol

SUMMARY:
The trial aims to investigate the effect of a topical application of a medical device based on inositol in recovering breast pain

DETAILED DESCRIPTION:
The present study enrolled patients with breast pain (measured through the VAS) aiming to evaluate the improvement of the pain after the local treatment

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 70 years
* Women who underwent breast surgery at least 15 days prior
* Women experiencing breast pain associated with the surgical wound

Exclusion Criteria:

* Women under the age of 18
* Ongoing systemic and/or local pain therapy
* Pregnant women

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female - breast pain
Enrollment: 50 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
Reduction of breast pain | 3 months
  Breast pain is evaluated by using VAS (Visual Analogue Scale)

SECONDARY OUTCOMES:
Follow up breast pain | 6 months
  Breast pain is evaluated by using VAS (Visual Analogue Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Umberto I, Roma, Italy

IPD SHARING:
Plan to Share IPD: No